CLINICAL TRIAL: NCT02041754
Title: Double Blind, Randomized, Placebo-controlled, Monocentric Clinical Investigation to Evaluate Efficacy of IQP-AK-102 on Appetite Reduction in Healthy Overweight and Obese Subjects
Brief Title: Safety and Efficacy of IQP-AK-102 in Reducing Appetite
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: InQpharm Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INQ/009913
Record Dates: First submitted 2014-01-19; First posted 2014-01-22 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Weight Loss; Appetite Modulation (Focus of Study)
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- IQP-AK-102 (Active Comparator): 2 capsules per dose, 3 times daily, 30-60 mins before each main meal with a full glass (250 mL) of water
  Interventions: Device: IQP-AK-102
- Placebo (Placebo Comparator): 2 capsules per dose, 3 times daily, 30-60 mins before each main meal with a full glass (250 mL) of water
  Interventions: Device: Placebo

INTERVENTIONS:
Device: IQP-AK-102
  Arms: IQP-AK-102
Device: Placebo
  Arms: Placebo

SUMMARY:
The individual ingredients in IQP-AK-102 have been widely used. Backed by data from several studies demonstrating their efficacy, we are conducting this study to look into the efficacy and safety of this novel combination of three fibres, in appetite regulation, aiming to reduce the appetite.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years
* 25≤BMI≤35
* Expressed desire for weight loss
* Accustomed to 3 main meals/day
* Generally in good health
* Consistent and stable body weight 3 months prior to study enrolment
* Consistent regular physical activity
* Commitment to avoid the use of other weight loss products during study
* Commitment to adhere to diet and lifestyle recommended for the study

Exclusion Criteria:

* Known sensitivity to the ingredients of the device
* Presence of any active gastrointestinal disease
* Malabsorption disorders
* Pancreatitis
* Stenosis in the GI tract
* Bariatric surgery
* Any other reason deemed suitable for exclusion, per investigator's judgement

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-01; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Difference of VAS between two study arms measured from time '0 to '240 during baseline visit and the final visit | 4 weeks
  Measured using a visual analogue scale (VAS)

SECONDARY OUTCOMES:
Difference in ad libitum energy intake between the two arms at baseline visit and at final visit | 4 weeks
  Measured in kcal
Change in "difference in ad libitum energy intake between two study arms", from baseline visit to the final visit | 4 weeks
  Measured in kcal
Difference in subjective appetite sensations (VAS) between baseline and the final visit for the two study arms | 4 weeks
  Measured using VAS
Difference in the mean change in body weight between the 2 arms, from baseline to the final visit | 4 weeks
  Measured in kg. Subjects wearing underwear and no shoes using calibrated weighing scales (Tanita BC-420 SMA)
Changes in waist and hip circumference | 4 weeks
  Measured in cm. Waist: measured at the level midway between the lateral lower rib margin and the iliac crest Hip: measured as the maximal circumference over the buttocks
Changes in body fat content and fat free mass | 4 weeks
  Measured in % and kg using bio-impedence method using validated electronic weighing scales (Tanita BC-420 SMA)
Subjects global feeling of satiety | 4 weeks
Food Craving Questionnaire | 4 weeks
  15 questions
Global evaluation of efficacy by the subjects and investigators | 4 weeks
Global evaluation of safety by the subjects and investigators | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Udo Bongartz, MD, Principal Investigator — Analyze & Realize
Locations (1):
- Udo Bongartz, Berlin, State of Berlin, Germany